CLINICAL TRIAL: NCT00031928
Title: Phase I Study of Intrathecal Mafosfamide
Brief Title: Mafosfamide in Treating Patients With Progressive or Refractory Meningeal Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000069240; NCI-90-C-0095K; BCM-H-3241
Record Dates: First submitted 2002-03-08; First posted 2003-01-27 (Estimated); Last update posted 2015-04-30 (Estimated); Status verified 2003-11

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: leptomeningeal metastases
MeSH Terms: conditions — Central Nervous System Neoplasms; Meningeal Carcinomatosis | interventions — mafosfamide

INTERVENTIONS:
Drug: mafosfamide

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase I trial to determine the effectiveness of mafosfamide in treating patients who have progressive or refractory meningeal tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the qualitative and quantitative toxicity of mafosfamide in patients with progressive or refractory meningeal malignancy.
* Determine the maximum tolerated dose of this drug in these patients.
* Determine the cerebrospinal fluid pharmacokinetics of this drug in these patients.

OUTLINE: This is a dose-escalation, multicenter study.

Patients receive intrathecal mafosfamide over 20 minutes twice weekly for 6 weeks (induction therapy). Patients then receive intrathecal mafosfamide once weekly for 4 weeks (consolidation therapy), twice a month for 4 months, and then monthly thereafter (maintenance therapy) in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of mafosfamide until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

PROJECTED ACCRUAL: A total of 3000 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of leukemia or lymphoma with meningeal involvement defined as cerebrospinal fluid cell count at least 5/mm^3 AND evidence of blast cells on cytospin preparation or by cytology OR
* Diagnosis of other solid tumor with meningeal involvement defined as presence of tumor cells on cytospin preparation or cytology OR presence of measurable meningeal disease on CT or MRI scan
* Meningeal malignancy must be progressive or refractory to conventional therapy

  * Meningeal malignancies secondary to an underlying solid tumor are allowed at initial diagnosis provided there is no conventional therapy
* No concurrent bone marrow relapse in leukemia or lymphoma patients
* No clinical evidence of obstructive hydrocephalus or compartmentalization of the cerebrospinal fluid flow as documented by a radioisotope indium In 111 or technetium Te 99-DTPA flow study

  * Patients demonstrating restored flow after focal radiotherapy are allowed

PATIENT CHARACTERISTICS:

Age:

* Over 3

Performance status:

* ECOG 0-2

Life expectancy:

* At least 8 weeks

Hematopoietic:

* Not specified

Hepatic:

* No clinically significant liver function abnormalities

Renal:

* No clinically significant renal function abnormalities

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 6 months after study
* No clinically significant metabolic parameter abnormalities (e.g., electrolytes, calcium, and phosphorus)
* No significant systemic illness (e.g., infection)

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Recovered from prior immunotherapy

Chemotherapy:

* At least 1 week since prior intrathecal chemotherapy (2 weeks for cytarabine (liposomal)) and recovered
* Concurrent systemic chemotherapy to control systemic or bulk CNS disease allowed with the following exceptions:

  * No phase I agent
  * No agent that significantly penetrates the CNS (e.g., high-dose systemic methotrexate (more than 1 g/m^2), high-dose cytarabine (more than 2 g/m^2), IV mercaptopurine, fluorouracil, topotecan, or thiotepa)
  * No agent known to have serious unpredictable CNS side effects

Endocrine therapy:

* Not specified

Radiotherapy:

* See Disease Characteristics
* Recovered from prior radiotherapy
* At least 8 weeks since prior craniospinal irradiation
* Local radiotherapy for symptomatic or bulky CNS disease must be given prior to induction therapy
* No concurrent whole brain or craniospinal irradiation

  * Concurrent partial brain (e.g., base of brain) or limited-field spinal radiotherapy for asymptomatic bulky (radiographically visible) CNS disease allowed
* Total CNS radiotherapy dose must not exceed accepted safe tissue tolerances

Surgery:

* Not specified

Other:

* At least 1 week since any prior CNS therapy
* At least 7 days since prior intrathecal investigational agent
* At least 14 days since prior systemic investigational agent
* No other concurrent intrathecal or systemic investigational agent
* No other concurrent intrathecal or systemic therapy to treat meningeal malignancy
* No other concurrent intrathecal therapy or agent that significantly penetrates the blood-brain barrier
* No concurrent agent known to have serious unpredictable CNS side effects

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3000 (Estimated)
Dates: Start 2002-01

CONTACTS AND LOCATIONS:
Overall Officials: Susan M. Blaney, MD, Study Chair — Texas Children's Cancer Center
Locations (9):
- United States (9):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Texas Children's Cancer Center, Houston, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Neurological Research Center, Inc., Bennington, Vermont
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington